CLINICAL TRIAL: NCT05566457
Title: Clinical Study of Huangshi Guizhi Wuwu Decoction in Improving the Paclitaxel-related Neurotoxicity in Breast Cancer Patients
Brief Title: HGWD Improve the Paclitaxel-related Neurotoxicity in Patients With BC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LQiao
Record Dates: First submitted 2022-09-14; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This open-label, single-center, prospective, randomized controlled trial was planned to be conducted in the National Cancer Center in China from January 2020 to June 2022.The eligible paticipants were assigned randomly in a 1:1 ratio to a study group (HGWD group) or a control group. PASS software (version 15.0) (Kaysville, Utah, USA) was used to calculate the sample size. Assuming α = 0.05 and 1-β = 0.8, a total of 80 patients were needed for the aim of decreasing the grade 2-3 PN from 60% to 30%. Assuming a lost-to-follow-up rate of 15%, a total of 92 patients were needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HGWD group (Experimental): Patients in the HGWD group (n = 46) soaked and washed Immersion and Washing limbs with HGWD infusion packs, followed by smearing limbs with vitamin E and vitamin B12. The composition of HGWD infusion pack was: 60g Radix Astragali (Huangqi), 15g Ramulus Cinnamomi (Guizhi), 15g Paeonia lactiflora (Baishao), 15g Gentiana (Qinjiao), 6g Scorpio (Quan-Xie), 20g Rhizoma Zingiberis Recens (Shengjiang), 20 Jujubes (Dazao), 30g Geranium wilfordii (Laoguancao), 12g radix sileris (Fangfeng), 30g Spatholobus suberectus (Jixueteng), 15g Ligusticum (Chuanxiong), 15g Poria (Fuling), and 15g Radixcyathulae (Chuanniuxi). HGWD infusion pack was boiled in water and extraction was performed twice to obtain a total of 500 ml drug-containing water. The drug-containing water was maintained at 39 to 40℃ for soaking and washing limbs for 20min twice a day for consecutive 14 days
  Interventions: Drug: Huangqi Guizhi Wuwu decoction (HGWD) infusion packs
- control group (Placebo Comparator): Patients in the control group and the HGWD group used vitamin E milk and vitamin B12 to smear the limbs three times per day for 14 days.
  Interventions: Drug: Huangqi Guizhi Wuwu decoction (HGWD) infusion packs

INTERVENTIONS:
Drug: Huangqi Guizhi Wuwu decoction (HGWD) infusion packs — Patients in the HGWD group (n = 46) soaked and washed Immersion and Washing limbs with HGWD infusion packs, followed by smearing limbs with vitamin E and vitamin B12. The composition of HGWD infusion pack was: 60g Radix Astragali (Huangqi), 15g Ramulus Cinnamomi (Guizhi), 15g Paeonia lactiflora (Baishao), 15g Gentiana (Qinjiao), 6g Scorpio (Quan-Xie), 20g Rhizoma Zingiberis Recens (Shengjiang), 20 Jujubes (Dazao), 30g Geranium wilfordii (Laoguancao), 12g radix sileris (Fangfeng), 30g Spatholobus suberectus (Jixueteng), 15g Ligusticum (Chuanxiong), 15g Poria (Fuling), and 15g Radixcyathulae (Chuanniuxi). HGWD infusion pack was boiled in water and extraction was performed twice to obtain a total of 500 ml drug-containing water. The drug-containing water was maintained at 39 to 40℃ for soaking and washing limbs for 20min twice a day for consecutive 14 days

SUMMARY:
The current treatments for albumin-bound paclitaxel (nab-PTX) -related peripheral neurotoxicity (PN) mainly included cryotherapy and compression therapy , oral B group vitamin , and duloxetine. However, treatment effectiveness of these three methods is limited. Huangqi Guizhi Wuwu decoction (HGWD) is an herbal formula recorded in "Synopsis of the Golden Chamber" for improving limb pain, tingling, and numbness, which is composed of five crude drugs (Astragali Radix, Cinnamomi Ramulus, Paeoniae Radix Alba, Zingiberis Rhizoma Recens, and Jujubae Fructus)(9). Recently, HGWD has been shown to be effective in the treatment of oxaliplatin- and diabetic-related PNs . But there are no prospective studies to explore the efficacy of HGWD in the treatment of nab-PTX-induced PN in patients with BC. Therefore, we conducted this prospective randomized controlled study to investigate the efficacy and safety of HGWD to prevent nab-PTX-induced PN in patients with BC. The primary aim of this study was to assess the prevention of nab-PTX-induced PN by soaking hands and/or feet with HGWD when compared to placebo.

DETAILED DESCRIPTION:
This open-label, single-center, prospective, randomized controlled trial was planned to be conducted in the National Cancer Center in China from January 2020 to June 2022.The eligible paticipants were assigned randomly in a 1:1 ratio to a study group (HGWD group) or a control group. PASS software (version 15.0) (Kaysville, Utah, USA) was used to calculate the sample size. Assuming α = 0.05 and 1-β = 0.8, a total of 80 patients were needed for the aim of decreasing the grade 2-3 PN from 60% to 30%. Assuming a lost-to-follow-up rate of 15%, a total of 92 patients were needed. The primary aim of this study was to assess the prevention of nab-PTX-induced PN by soaking hands and/or feet with HGWD when compared to placebo.

ELIGIBILITY:
The inclusion criteria comprised:

ˑ histologically confirmed untreated BC; ˑ female; ˑage from 18 to 65 years old; ( ˑ Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1; ˑat least receiving 4 cycles of nab-PTX (260mg/m2); ˑ grade 2 or greater nab-PTX induced-PN evaluated by European Organisation for the Research and Treatment of Cancer-Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20)(12, 13); ˑ estimated survival time > 6 months. The exclusion criteria were： ˑ a history of diabetes or neurological disorders; ˑmental disorder; ˑabnormal hepatic functions (total bilirubin upper limit of normal (ULN), alanine transaminase/aspartate transaminase ≥ 2.5 × ULN ), renal functions(creatinine ≥ 1.5 × ULN), and hematological functions (absolute neutrophil count ≤ 1.5 × 109/L, platelet count ≤ 80 × 109/L, hemoglobin < 90 g/L); ˑFailure to complete chemotherapy due to treatment-related adverse events; ˑ a family history of a genetic neuropathy; ˑhad received previous treatment with neurotoxic chemotherapy, including oxaliplatin, cisplatin, vinca alkaloid and etc.; ˑ a history of allergy to Chinese medicine.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
European Organisation for the Research and Treatment of Cancer-Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20) questionnaire | up to 3 months
  The primary outcome measures was European Organisation for the Research and Treatment of Cancer-Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20) questionnaire, which consisted of 20 items that graded the degree of functioning affected by sensory (9 items), motor (8 items) and autonomic CIPN symptoms (3 items). Each item was scored from 1 to 4 (corresponding to answers of none, mild, moderate, and severe) on a Likert scale and subsequently the scores were summed up (total score range, 1-44). Sensory raw scale scores range from 1 to 36, motor raw scale scores range from 1 to 32, and autonomic raw scale scores range from 1 to 12 for men and 1-8 for women (erectile function item is excluded). Higher scores represented more symptoms and worse quality of life.

SECONDARY OUTCOMES:
European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) (version 3) | up to 3 months
  The EORTC QLQ-C30 is a validated 30-item questionnaire containing both single- and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality of Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). Scores for each scale and single-item measure are averaged and transformed linearly to a score ranging from 0-100. A high score for functional scales and for Global Health Status/QoL represent better functioning ability or HRQoL, whereas a high score for symptom scales and single items represents significant symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, Dr., Principal Investigator — Department of Medical Oncology, National Cancer Center
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No